CLINICAL TRIAL: NCT05840614
Title: The Effectiveness of a Remote Family Support Programs for Families of Patients With Eating Disorders
Brief Title: The Remote Family Support Programs for Eating Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nagoya City University (Other)
Responsible Party: Principal Investigator, Fujika Katsuki, Professor, Nagoya City University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NagoyaCU
Record Dates: First submitted 2023-04-21; First posted 2023-05-03 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Eating Disorders
Keywords: Family support, Interpersonal psychotherapy
MeSH Terms: conditions — Feeding and Eating Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- The remote family support program plus TAU (Experimental): Behavioral: The remote family support program Remote family support programs consist of interpersonal psychotherapy (IPT) and family psychoeducation.
  Interventions: Behavioral: The remote family support program
- Treatment as Usual (No Intervention): Treatment as usual administrated by physician.

INTERVENTIONS:
Behavioral: The remote family support program — Remote family support programs consist of interpersonal psychotherapy (IPT) and family psychoeducation.
  Each session consisted of a lecture, followed by role playing and supportive group therapy. In the first session, we informed the participants about the symptoms of eating disorders and mechanism of IPT; in the second session, we shared details about the characteristics of adolescents; and during the third and fourth sessions, we provided information on effective communication according to IPT.
  Arms: The remote family support program plus TAU

SUMMARY:
Eating disorders are serious mental health disorders associated with high levels of mortality, disability, physical and psychological morbidity, and impaired quality of life. Family members who spend the majority of their time with patients of eating disorders experience heavy psychological burden. Remote family support programs consist of interpersonal psychotherapy and family psychoeducation. This study aimed to examine the effectiveness of a remote family support program for eating disorders in an RCT (randomized controlled trial). The specific objective was to conduct a small pilot RCT of the remote family support program (n=28) compared with TAU (n=28).

ELIGIBILITY:
Inclusion Criteria:

* The research participants are parents of patients who have been diagnosed with an eating disorder by a physician or have symptoms of an eating disorder; parents may or may not be related by blood.
* The ABOS score measured by the research participants at enrollment is over 8 points.
* Patient age at enrollment ranged from 12 to 29 years.
* The patient has lived with their parents at the time of participating in this study and is expected to live with them during the investigation period.
* Patients may or may not undergo treatment.
* Patients with other psychiatric comorbidities are included.
* Participants with other psychiatric comorbidities are included.
* If multiple family members (e.g., parents) participated in this program, the primary participant is determined, and that person becomes the target research participant.
* Willingness to provide informed consent and comply with the trial protocol.

Exclusion Criteria:

* The participants cannot read or write in Japanese
* The participants cannot use the Zoom meeting system
* Researcher of this study and their families

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2023-03-18 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
Change in the total Active Listening Attitude Scale (ALAS) score of participants | Base-line, four weeks, and eight weeks
  The ALAS comprises 2 subscales and 20 items: listening attitude (10 items) and listening skills (10 items). Higher the scores indicate better listening attitudes or skills.

SECONDARY OUTCOMES:
Change in the total Social Provisions Scale-10 item (SPS-10) score of participants | Base-line, four weeks, and eight weeks
  Parents' perception of social support is measured using SPS-10.

OTHER OUTCOMES:
Loneliness | Base-line, four weeks, and eight weeks
  Parents' loneliness is evaluated using the University of California Los Angeles Loneliness Scale (ULS).
Mental health | Base-line, four weeks, and eight weeks
  Psychological distress experienced by the participants is assessed using the Kessler Psychological Distress Scale (K6).
Family functioning | Base-line, four weeks, and eight weeks
  Family functioning is assessed using the Family Assessment Device (FAD).
Eating disorder behaviors | Base-line, four weeks, and eight weeks
  Information on behaviors and attitudes of patients with eating disorders obtained from their parents is measured using the Anorectic Behavior Observation Scale (ABOS).

CONTACTS AND LOCATIONS:
Overall Officials: Fujika Katsuki, Ph.D., Principal Investigator — Nagoya City University
Locations (1):
- Fujika Katsuki, Nagoya, Aichi-ken, Japan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Katsuki F, Sawada H, Kawasaki Y, Kondo M, Yamada A, Watanabe N. Effectiveness of Remote Family Education and Support Program for Parents of Adolescents With Eating Disorders Based on Interpersonal Psychotherapy: A Randomized Controlled Trial. Int J Eat Disord. 2025 Dec;58(12):2281-2291. doi: 10.1002/eat.24541. Epub 2025 Sep 3. PMID 40899790
- [Derived] Katsuki F, Watanabe N, Kondo M, Sawada H, Yamada A. Remote family education and support program for parents of patients with adolescent and early adulthood eating disorders based on interpersonal psychotherapy: study protocol for a pilot randomized controlled trial. J Eat Disord. 2024 May 17;12(1):61. doi: 10.1186/s40337-024-01013-z. PMID 38760800
- See also: Fujika Katsuki, et. al.: Remote family education and support program for parents of patients with adolescent and early adulthood eating disorders based on interpersonal psychotherapy: study protocol for a pilot randomized controlled trial — https://jeatdisord.biomedcentral.com/articles/10.1186/s40337-024-01013-z